CLINICAL TRIAL: NCT03912688
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Remifentanil Consumption and Postoperative Pain in Patients Undergoing Radical Mastectomy
Brief Title: TEAS Reduces Remifentanil Consumption
Acronym: TRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, principle investigator, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJA-S-20190212
Record Dates: First submitted 2019-02-12; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Acupuncture Points

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Interventions were performed by a designated investigator who was not involved in the anaesthesia or the follow-up. The stimulator was placed in an opaque box to blind the surgical team and the anesthesiologists to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single acupoint stimulation (Experimental)
  Interventions: Device: acupoint stimulation; Device: single acupoint
- dual acupoints stimulation (Experimental)
  Interventions: Device: acupoint stimulation; Device: dual acupoints
- no stimulation (No Intervention)

INTERVENTIONS:
Device: acupoint stimulation
  Arms: dual acupoints stimulation; single acupoint stimulation
Device: single acupoint
  Arms: single acupoint stimulation
Device: dual acupoints
  Arms: dual acupoints stimulation

SUMMARY:
Transcutaneous electrical acupoint stimulation (TEAS) has been shown to decrease the need of opioids including remifentanil during anaesthesia. However, it is not clear whether combination of two or more acupoints could induce stronger analgesia. Moreover, evidence for the long-term effect of TEAS has been limited. The present study was to compare the short-term and long-term effect on pain of dual-acupoint and single-acupoint TEAS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 yrs
* body mass index (BMI) of 18 to 30 kg/m2
* elective radical mastectomy under general anaesthesia

Exclusion Criteria:

* contradictions to TEAS
* difficulties in communication
* histories of general anaesthesia
* drug or alcohol abuse or addiction
* cardiac dysfunction or severe hypertension
* confirmed hepatic dysfunction and renal impairment
* the participants recruited into other clinical trials during last three months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
consumption of remifentanil | from start of anesthesia to extubation, on average 2 hours

SECONDARY OUTCOMES:
time to recall | from end of remifentanil infusion to patient response to verbal command,approximately 10 minutes on average
time to extubation | from end of remifentanil infusion to extubation,approximately 10 minutes on average
respiratory depression | end of the surgery to discharge from postanesthesia care unit,with an average of 30 minutes
nausea and vomiting | end of the surgery to discharge from postanesthesia care unit,with an average of 30 minutes
visual analogue scale of pain | end of the surgery to discharge from postanesthesia care unit,with an average of 30 minutes
  pain intensity is assessed by a 0-10mm scale, 0 is no pain, 10 is untolerated pain
patients' satisfaction score | from end of surgery to 24 hours after surgery, totally 24 hours
  patients' satisfaction score is assessed by a 0-10mm scale, 0 is no pain, 10 is untolerated pain
incidence of pain at 3m after surgery | from discharge from hospital to 3 months after surgery, approximately 3 months
  percentage of patients suffering from pain around the incision
incidence of pain at 6m after surgery | from discharge from hospital to 6 months after surgery, approximately 3 months
  percentage of patients suffering from pain around the incision

REFERENCES:
- [Background] Kuhn LA. Editorial: Acupuncture anesthesia for open heart surgery. Am J Cardiol. 1974 Aug;34(2):254-5. doi: 10.1016/0002-9149(74)90207-0. No abstract available. PMID 4843161
- [Result] Lu Z, Dong H, Wang Q, Xiong L. Perioperative acupuncture modulation: more than anaesthesia. Br J Anaesth. 2015 Aug;115(2):183-93. doi: 10.1093/bja/aev227. PMID 26170347
- [Result] Wang H, Xie Y, Zhang Q, Xu N, Zhong H, Dong H, Liu L, Jiang T, Wang Q, Xiong L. Transcutaneous electric acupoint stimulation reduces intra-operative remifentanil consumption and alleviates postoperative side-effects in patients undergoing sinusotomy: a prospective, randomized, placebo-controlled trial. Br J Anaesth. 2014 Jun;112(6):1075-82. doi: 10.1093/bja/aeu001. Epub 2014 Feb 26. PMID 24576720
- [Result] Yan B, Li K, Xu J, Wang W, Li K, Liu H, Shan B, Tang X. Acupoint-specific fMRI patterns in human brain. Neurosci Lett. 2005 Aug 5;383(3):236-40. doi: 10.1016/j.neulet.2005.04.021. PMID 15876491